CLINICAL TRIAL: NCT05423535
Title: A Randomized Controlled Trial Comparing Hemostatic Gelatin Sponge to Collagen Matrix as Socket Seal in Alveolar Ridge Preservation
Brief Title: Hemostatic Gelatin Sponge Versus Collagen Matrix in Alveolar Ridge Preservation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants Enrolled
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BC-11345
Record Dates: First submitted 2022-06-03; First posted 2022-06-21 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Changes in Soft Tissue Height

STUDY DESIGN:
Intervention Model Description: Intra-subject RCT with 2 treatment arms (control group: collagen matrix; test group: hemostatic gelatine sponge). In every patient two teeth are extracted. Coincidence (coin flip) will determine which site is treated with the gelatine sponge and which with the collagen matrix.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: It concerns a surgical intervention. Hence, the treating surgeon cannot be masked. As each patient receives both the control and test treatment at the same moment, the patient is masked. The investigators and outcome assessors are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: Collagen Matrix (Active Comparator): collagen matrix: Mucograft Seal®, Geistlich Pharma AG, Wolhusen, Switzerland
  Interventions: Device: test group: collagen matrix (Mucograft Seal®, Geistlich Pharma AG, Wolhusen, Switzerland)
- Test group: Hemostatic Gelatin Sponge (Experimental): Hemostatic gelatin spons: Spongostan Dental® 1x1x1 cm, Ethicon, Johnson & Johnson, New Brunswick, VS
  Interventions: Device: test group: collagen matrix (Mucograft Seal®, Geistlich Pharma AG, Wolhusen, Switzerland)

INTERVENTIONS:
Device: test group: collagen matrix (Mucograft Seal®, Geistlich Pharma AG, Wolhusen, Switzerland) — Following tooth extraction and wound debridement, the alveolar socket was filled with collagen-enriched deproteinized bovine bone mineral (C-DBBM, Bio-Oss Collagen® 100 mg or 250 mg, Geistlich Pharma AG, Wolhusen, Switzerland) up to the level of the oral bone crest. Subsequently, a collagen matrix (Mucograft Seal®, Geistlich Pharma AG, Wolhusen, Switzerland) or gelatin spons (Spongostan Dental® 1x1x1 cm, Ethicon, Johnson & Johnson, New Brunswick, VS) was sutured on top with 4 to 6 single sutures (Seralon 6/0, Serag Weissner, Naila, Germany) to protect the underlying C-DBBM.
  Other Names: control group: gelatin spons (Spongostan Dental® 1x1x1 cm, Ethicon, Johnson & Johnson, New Brunswick, VS)

SUMMARY:
Patients in need of extraction of two teeth followed by implant replacement, with > 50% buccal bone present following tooth extraction and with 1 or 2 neighbouring teeth present, were invited to participate in an intra-subject RCT comparing hemostatic gelatin sponge to collagen matrix as socket seal in alveolar ridge preservation.

The sample size calculation indicated 16 patients to be included per group. To compensate for dropouts, this number was increased to 20 patients per group. Coincidence (coin flip) determined which site is treated with the gelatine sponge and which with the collagen matrix.

Teeth were extracted without flap elevation. When deemed necessary by the clinician, papillary incisions were made for minimal reflection, which enabled to place elevators without damaging soft tissues. Buccal soft tissues were never raised. Following wound debridement and rinsing, the alveolar socket was filled with collagen-enriched deproteinized bovine bone mineral (C-DBBM, Bio-Oss Collagen® 100 mg or 250 mg, Geistlich Pharma AG, Wolhusen, Switzerland) up to the level of the oral bone crest. Subsequently, a collagen matrix (Mucograft Seal®, Geistlich Pharma AG, Wolhusen, Switzerland) or gelatin spons (Spongostan Dental® 1x1x1 cm, Ethicon, Johnson & Johnson, New Brunswick, VS) was sutured on top with 4 to 6 single sutures (Seralon 6/0, Serag Weissner, Naila, Germany) to protect the underlying C-DBBM.

Changes in soft tissue height at the buccal and oral aspect is the primary outcome. A small-field low-dose CBCT image was taken at T0 (immediately postop) and T3 (4 months). Those images were superimposed in specialized software (OnDemand3D, Cybermed Inc., Seoul, South-Korea). Changes in soft tissue height were calculated by subtracting soft tissue height at T3 from soft tissue height at T0.

Secondary outcomes included wound healing and closure in the first three weeks, changes in hard and soft tissues and mucosal scarring after 4 months.

ELIGIBILITY:
Inclusion Criteria:

* good oral hygiene (plaque score < 25%)
* 1 or 2 neighbouring teeth present
* in need for extraction of two teeth, followed by implant placement
* >50% bone present
* signed informed consent

Exclusion Criteria:

* systematic diseases
* smoking
* history of periodontitis
* untreated caries lesions
* pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-06 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in soft tissue height at the buccal and lingual aspect | T0 (immediately post-op) and T3 (4 months)
  A CBCT was taken at T0 (immediately post-op) and T3 (4 months). Since soft tissues were separated from hard tissues by using lip retractors and a backward position of the tongue, soft tissue height could be assessed on CBCT images. Changes in soft tissue height were calculated by subtracting soft tissue height at T3 from soft tissue height at T0.

SECONDARY OUTCOMES:
Wound healing | T1 (1 week), T2 (3 weeks) and T3 (4 months)
  Socket wound healing score (SWHS). SWHS was assessed on the basis of occlusal clinical pictures and results in the following scores: 0 = Wound covered with keratinized gingiva, pink tissue color, no bleeding, continuous with healthy tissue; 1 = Socket filled with organized granulation tissue, no bleeding, collapsed to a depth of 0 - 2 mm from the buccal gingival margin; 2 = Socket filled with organized granulation tissue, ¼ to ½ of the wound showing red tissue color, no bleeding, collapsed to a depth of 2 - 4 mm from the buccal gingival margin; 3 = Socket filled with unorganized granulation tissue, more than ½ of the wound showing red tissue color, bleeding, no evidence of acute infection; 4 = Socket is filled with foreign material (food, etc.) and shows signs of alveolitis.
  The higher the score, the worser the outcome.
Wound dimension | T0 (immediately post-op), T1 (1 week) and T3 (4 months)
  Bucco-lingual and mesio-distal wound dimensions were registered with a periodontal probe to the nearest 0.5 mm at T0 (immediately postop), T1 (1 week) and T3 (4 months).
Changes in buccal soft tissue profile | T0 (immediately post-op) and T3 (4 months)
  An intra-oral scan was taken at T0 (immediately postop) and T3 (4 months). The obtained digital surface models in STL format were imported into designated software to analyze profilometric changes. A study-relevant area of interest (AOI) at the buccal aspect was selected for each site. The AOI varied between sites due to individual anatomic differences but was kept constant in each site across timepoints. Digital surface models were superimposing using the best-fit algorithm at the unchanged adjacent tooth surfaces. A mean volumetric change (mm3) within the AOI for each site from T0 to T3 was calculated by the software and divided by the AOI resulting in a mean change in buccal soft tissue profile. Details on the method can be found in an earlier paper (Eeckhout et al., 2020).
Mucosal scarring | T3 (4 months)
  The Mucosal Scarring Index (MSI) (Wessels et al., 2019) was registered on the basis of frontal and occlusal clinical pictures. The MSI results in a score from 0 (no scar) to 10 (most extreme scar).
  The higher the score, the worser the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Cosyn, Professor, Principal Investigator — University Ghent
Locations (2):
- Belgium (2):
  - BV Paro Glibert, Geraardsbergen, Oost-Vlaanderen
  - Centrum voor Parodontologie en Orale Implantologie, Zottegem, Oost-Vlaanderen